CLINICAL TRIAL: NCT02801773
Title: Clinical Effect of Lactobacillus Reuteri in Treatment of Gingivitis. Randomized Clinical Trials
Brief Title: Clinical Effect of Lactobacillus Reuteri in Treatment of Gingivitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Jorge Gamonal, Proffesor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1130570-Fondecyt
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Gingivitis
Keywords: gingivitis; probiotic; non- surgical treatment
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Gingivitis with Probiotic (Experimental): Gingivitis group of patient treated with conventional therapy (scaling, coronary polish and oral higiene instruction) and adjunct probiotic one lozenge containig Lactobacillus reuteri per day during 3 month
  Interventions: Dietary Supplement: Treatment Gingivitis with Probiotic
- Treatment Gingivitis conventional (Placebo Comparator): Gingivitis group of patient treated with conventional therapy (scaling, coronary polish and oral higiene instruction) and one lozenge containig placebo (mint lozenge) per day during 3 month
  Interventions: Other: Treatment Gingivitis conventional

INTERVENTIONS:
Dietary Supplement: Treatment Gingivitis with Probiotic — Gingivitis Treatment (scaling and coronary polish) and one lozenge containing Lactobacillus reuteri per day during 3 months
  Arms: Treatment Gingivitis with Probiotic
Other: Treatment Gingivitis conventional — gingivis treatment (scaling and coronary polish) and and one lozenge containing Placebo (mint lozenge) per day during 3 months
  Arms: Treatment Gingivitis conventional

SUMMARY:
The aim of this randomized placebo- controlled clinical trials is to evaluate the effects of Lactobacillus reuteri containing probiotic lozenges as an adjunct to scaling and root planning (SRP). Material and methods: Thirty six gingivitis patients will be recruited and monitored clinically at baseline, 3 and 6 month after therapy. All patients will receive scaling and periodontal treatment and randomly will be assigned over an experimental (SRP + probiotic, N=18) or control (SRP+ placebo, n=18) group. The lozenges will be used once per day during 3 month.

DETAILED DESCRIPTION:
Gingivitis is the most prevalent worldwide periodontal disease, is characterized by inflammation of the tissues surrounding the tooth without causing periodontal attachment loss. Preventive and / or therapeutic measures to facilitate or improve their control are therefore very important, much more if you consider that gingivitis and periodontitis are considered part of an ongoing inflammatory process. Treatment of gingivitis, like that of all periodontal diseases has been based on the implementation of control measures personal and professional plaque. Notwithstanding the foregoing, it has been reported that although mechanical therapy achieved significantly decrease the periodontopathogens, this may be only temporary since bacteria can recolonize the treated niches in the oral cavity. In this context, it has emerged as a new treatment strategy complementary use of probiotics such as Lactobacillus reuteri, which possess anti-bacterial and anti-inflammatory properties. Generally speaking, probiotics would promote health by competitive exclusion of some or positive pathogenic bacteria. Objective: To evaluate the effect of the administration of Lactobacillus reuteri as an adjunct to conventional periodontal therapy in adolescent and young adult patients with gingivitis. Methodology: A randomized double-blind clinical trial to evaluate the effect of probiotic lozenges Lactobacillus rhamnosus as an adjunct to conventional periodontal treatment of patients with gingivitis will be performed. Expected Results: Statistically significant decrease in bleeding and gingival index in the experimental group compared with the control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gingivitis
* Gingival index > 1.5 (> 10 % of sites examined)
* Bleeding index > 10 % sites surveyed
* Probing Depth < 4 mm
* Systemically healthy (except for the presence of gingivitis)
* Patients who have not received periodontal treatment before the test and no intake of medicines such antibiotic and/ or anti-inflammatory in the last 3 months prior to the start of the study

Exclusion Criteria:

* Patient who develop systemic disease during the study
* Patient who have to ingest antibiotic/ or anti-inflammatories during the study
* If you are a woman becomes pregnant during the study

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Differences between groups for bleeding on probing changes | baseline, 1, 3 month

SECONDARY OUTCOMES:
Differences between groups for gingival index | baseline, 1, 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gamonal Aravena, Proffesor, Principal Investigator — Faculty of Dentistry of University of Chile
Locations (1):
- Faculty of Dentistry of University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No